CLINICAL TRIAL: NCT02702765
Title: Macrophages and the Macrophage Activation Markers sCD163 and Mannose Receptor (sMR) in Patients With Wilsons Disease - Associations With Liver Disease Severity and Fibrosis
Brief Title: sCD163 and sMR in Wilsons Disease - Associations With Disease Severity and Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Wilson sCD163
Record Dates: First submitted 2016-02-26; First posted 2016-03-09 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Wilsons Disease
Keywords: sCD163; liver cirrhosis; disease severity
MeSH Terms: conditions — Hepatolenticular Degeneration; Liver Cirrhosis | interventions — High-Energy Shock Waves; Galactose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Wilsons disease (Experimental): All patients will receive all interventions (galactose elimination capacity test , ultrasound, fibroscan, continuous reaction time test and functional hepatic nitrogen clearance ), except liver biopsy.
  Interventions: Procedure: Fibroscan; Procedure: Ultrasound; Drug: Galactose; Procedure: Liver biopsy; Procedure: Functional hepatic nitrogen clearance

INTERVENTIONS:
Procedure: Fibroscan — Liver fibrosis will be determined using fibroscan, and reported as changes in the amount of fibrosis in the liver. The fibroscan is a non-invasive procedure
Procedure: Ultrasound — Ultrasound is a non-invasive procedure
Drug: Galactose — Galactose elimination capacity is performed to evaluate metabolic liver function.
  The metabolic liver function test galactose elimination capacity requires a 6-hour fast, the infusion of galactose, blood sampling from the ear lobe, and collection of urine for 4 hours.
  Other Names: Galactose elimination capacity
Procedure: Liver biopsy — Histological disease activity at time of diagnosis evaluating if any liver fibrosis
Procedure: Functional hepatic nitrogen clearance — Functional hepatic nitrogen clearance to evaluate metabolic liver function Functional hepatic nitrogen clearance requires a 12-hour fast, two venflons, the infusion of alanine, and urine sampling for 4 hours

SUMMARY:
The aim is to investigate macrophage activation markers and correlations to liver fibrosis in patients with Wilsons Disease. Researchers wish to investigate associations to neurologic and metabolic liver function. Researchers will assess this by comparing blood samples with fibrosis and liver function analyses. This study provides new insight into macrophages and their involvement in Wilsons Disease.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Wilsons disease

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Measurement of the macrophage activation markers sCD163 | Baseline, 1 year, 2 year, 3 year
  For the investigations a total of 100 ml of blood is drawn, all stored in a research biobank.
Measurement of soluble mannose receptor (sMR) | Baseline, 1 year, 2 year, 3 year
  For the investigations a total of 100 ml of blood is drawn, all stored in a research biobank.

SECONDARY OUTCOMES:
Urinary copper excretion in 24 hour urine collection | Baseline, 1 year, 2 year, 3 year
  The patient collects urine for 24 hours at home in a designated container, which is handed out at the department. The container is kept refrigerated and is brought to the control
Ultrasound is performed for signs of liver cirrhosis. | Baseline, 1 year, 2 year, 3 year
  Ultrasound is a non-invasive procedure. Signs og liver cirrhosis by ultrasound are surface modularity, a smaller liver, heterogeneous echo texture and signs of portal hypertension.
Fibroscan is performed to evaluate liver stiffness (fibrosis) | Baseline, 1 year, 2 year, 3 year
  Liver fibrosis will be determined using fibroscan, and reported as changes in the amount of fibrosis in the liver. The fibroscan is a non-invasive procedure.
Continous Reaction Time to evaluate brain dysfunction | Baseline, 1 year, 2 year, 3 year
  Continous Reaction Time is a computerized 10 minutes test that measures and combines motor reaction speed and sustained attention.
Galactose elimination capacity is performed to evaluate metabolic liver function | Baseline, 1 year, 2 year, 3 year
  The metabolic liver function test Galactose elimination capacity requires a 6-hour fast, the infusion of galactose, blood sampling from the ear lobe, and collection of urine for 4 hours.
Histological disease activity at time of diagnosis and liver biopsy, evaluating if any liver fibrosis | Baseline, 1 year, 2 year, 3 year
  Liver fibrosis will be also be determined on liver biopsies.
Functional hepatic nitrogen clearance to evaluate metabolic liver function | Baseline, 1 year, 2 year, 3 year
  Functional hepatic nitrogen clearancerequires a 12-hour fast, two venflons, the infusion of alanine, and urine sampling for 4 hours. It evaluates the metabolic liver function by measuring the clearance of alanine from blod by analyzing the amount og urea in the urine collected 4 hours after the start og the alanine infusion.
The Portosystemic Encephalopathy to evaluate brain dysfunction | Baseline, 1 year, 2 year, 3 year
  The Portosystemic Encephalopathy test is a 15-minute paper-pencil test battery comprised of 5 sub-tests: Digit Symbol test (DST), Number Connection Test A (NCT-A), Number Connection Test B (NCT-B), Serial Dotting Test (SDOT), and Line Tracing Test (LTT, time and errors).

CONTACTS AND LOCATIONS:
Overall Officials: Henning Grønbæk, Professor, Principal Investigator — Aarhus University Hospital, Nørrebrogade 44, Aarhus C, Denmark, 8000
Locations (1):
- Department of Hepatology and Gastroenterology, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Bjorklund J, Laursen TL, Sandahl TD, Moller HJ, Vilstrup H, Ott P, Gronbaek H. High hepatic macrophage activation and low liver function in stable Wilson patients - a Danish cross-sectional study. Orphanet J Rare Dis. 2018 Sep 21;13(1):169. doi: 10.1186/s13023-018-0910-7. PMID 30241550